CLINICAL TRIAL: NCT07138144
Title: Efficacy, Safety, and Tolerability of Switching to a Two-Drug Regimen With DTG/3TC Compared to Maintaining a Three-Drug Regimen With BIC/FTC/TAF or DTG/3TC/ABC in Virologically Suppressed PeopLe Living With HIV After 24 and 48 Weeks of Follow-Up
Acronym: TLACAELEL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: José Antonio Mata Marín (Other Government)
Responsible Party: Sponsor-Investigator, José Antonio Mata Marín, Doctor, Instituto Mexicano del Seguro Social
Organization: Instituto Mexicano del Seguro Social (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2025-3502-186
Record Dates: First submitted 2025-08-04; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: HIV Infections
Keywords: HIV; DTG/3TC; BIC/TAF/FTC; dual therapy; non-inferiority
MeSH Terms: conditions — HIV Infections | interventions — Dual Anti-Platelet Therapy

STUDY DESIGN:
Intervention Model Description: This is a phase 4, randomized, controlled, open-label, single-center clinical trial conducted at the Hospital de Infectología, National Medical Center "La Raza." The study employs a non-inferiority design with follow-up assessments at 24 and 48 weeks. The study will enroll 156 PLWH aged ≥18 years who are on ART with BIC/FTC/TAF or DTG/3TC/ABC and have maintained virological suppression (HIV-1 RNA <50 copies/mL) for at least 48 weeks. Participants will be randomized in a 2:1 ratio: 104 to switch to DTG/3TC and 52 to continue their current regimen (control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standar therapy (Active Comparator): Bictegravir 50 mg / tenofovir alafenamide 25 mg / emtricitabine 200 mg or dolutegravir 50 mg / lamivudine 300 mg / abacavir 600 mg, both combinations in a single tablet, will be used as standard therapy
  Interventions: Drug: Standard Medical Therapy
- dual therapy (Experimental): This arm is the experimental one, with dual therapy, 2 drugs: Dolutegravir 50 mg/Lamivudina 300 mg, in a single tablet.
  Interventions: Drug: dual therapy

INTERVENTIONS:
Drug: Standard Medical Therapy — Intervention arm will be dual therapy oh DTG 50 mg/ 3TC 300 mg, this will be compared to standar therapy of 3 drugs with: Bictegravir 50 mg / tenofovir alafenamide 25 mg / emtricitabine 200 mg or dolutegravir 50 mg / lamivudine 300 mg / abacavir 600 mg, both combinations in a single tablet.
  Other Names: INSTI
  Arms: Standar therapy
Drug: dual therapy — Intervention arm will be dual therapy oh DTG 50 mg/ 3TC 300 mg, this will be compared to standar therapy of 3 drugs
  Other Names: DTG/3TC
  Arms: dual therapy

SUMMARY:
This is a phase 4, randomized, controlled, open-label, single-center clinical trial conducted at the Hospital de Infectología, National Medical Center "La Raza." The study employs a non-inferiority design with follow-up assessments at 24 and 48 weeks. The study will enroll 156 PLWH aged ≥18 years who are on ART with BIC/FTC/TAF or DTG/3TC/ABC and have maintained virological suppression (HIV-1 RNA <50 copies/mL) for at least 48 weeks. Participants will be randomized in a 2:1 ratio: 104 to switch to DTG/3TC and 52 to continue their current regimen (control group).

DETAILED DESCRIPTION:
Since the identification of the human immunodeficiency virus (HIV), developing effective, safe, and well-tolerated antiretroviral therapy (ART) for people living with HIV (PLWH) has been a global health priority. Advances in ART have significantly improved the prognosis for PLWH, achieving life expectancies comparable to the general population. However, three-drug regimens, such as bictegravir/emtricitabine/tenofovir alafenamide (BIC/FTC/TAF) or dolutegravir/lamivudine/abacavir (DTG/3TC/ABC), are associated with metabolic, renal, and cardiovascular adverse effects, particularly in the Mexican population, which has a high prevalence of metabolic syndrome.

Clinical trials, including GEMINI, TANGO, SALSA, RUMBA, PASO DOBLE, and DYAD, have demonstrated that two-drug regimens, such as dolutegravir/lamivudine (DTG/3TC), offer comparable virological efficacy and improved tolerability. Reducing the pharmacological burden may minimize adverse effects while maintaining viral suppression. The impact of metabolic disturbances on fat weight gain remains a controversial issue.

Objectives General Objective To compare the effectiveness, safety, and tolerability of switching to a DTG/3TC regimen versus continuing BIC/FTC/TAF or DTG/3TC/ABC in virally suppressed PLWH at 24 and 48 weeks of treatment.

Secondary Objectives

* Assess changes in lipid profile, body mass index (BMI), and abdominal circumference.
* Evaluate alterations in glucose metabolism.
* Measure changes in blood pressure and cardiovascular risk using Framingham and AHA/ACC scales.
* Analyze changes in body composition (fat, water, muscle).
* Document adverse events associated with ART. Study Design This is a phase 4, randomized, controlled, open-label, single-center clinical trial conducted at the Hospital de Infectología, National Medical Center "La Raza." The study employs a non-inferiority design with follow-up assessments at 24 and 48 weeks. The study will enroll 156 PLWH aged ≥18 years who are on ART with BIC/FTC/TAF or DTG/3TC/ABC and have maintained virological suppression (HIV-1 RNA <50 copies/mL) for at least 48 weeks. Participants will be randomized in a 2:1 ratio: 104 to switch to DTG/3TC and 52 to continue their current regimen (control group).

Inclusion Criteria

* Age ≥18 years.
* Virological suppression (HIV-1 RNA <50 copies/mL) for ≥48 weeks.
* Estimated glomerular filtration rate (eGFR) ≥60 mL/min.
* Signed informed consent. Exclusion Criteria
* Pregnancy or breastfeeding.
* Hepatitis B or C coinfection.
* Active malignancy.
* Use of recreational drugs or medications with significant interactions with ART.

Procedures Following approval by the local ethics committee, participant recruitment will commence. Participants will be followed continuously for 48 weeks. Data will be collected on efficacy (viral suppression), safety (adverse events), and tolerability (patient-reported outcomes and clinical assessments).

Data Management and Statistical Analysis

Patient data will remain confidential and accessible only to study investigators. Data will be recorded in an SPSS database. Statistical analyses will include:

* Kolmogorov-Smirnov test for normality.
* χ² test for categorical variables.
* Student's t-test or Mann-Whitney U test for continuous variables, as appropriate.
* ANOVA for group comparisons.
* Paired tests for within-group changes. A significance level of p ≤ 0.05 will be applied.

Feasibility The Hospital de Infectología, National Medical Center "La Raza," has the necessary infrastructure, trained personnel, and access to study medications to conduct this trial. The study is independent and not sponsored by any pharmaceutical company.

ELIGIBILITY:
Inclusion Criteria:

* PLWH aged over 18 years.
* Virologically suppressed for at least 48 weeks prior to study enrollment.
* On ART with Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/FTC/TAF) or Dolutegravir/Lamivudine/Abacavir (DTG/3TC/ABC).
* No history of virologic failure.
* Willing to participate in the study.
* Signed written informed consent.
* HIV-1 RNA <50 copies/mL within 4 weeks prior to randomization.
* eGFR by CKD-EPI ≥60 mL/min.

Exclusion Criteria:

* Pregnant or breastfeeding patients.
* Known allergies to any component of the antiretroviral regimens.
* Coinfection with hepatitis B and/or hepatitis C virus.
* Concomitant medications that interact with any component of the ART regimens.
* Diagnosis of malignancy prior to randomization.
* Use of recreational drugs with anorexigenic potential (crystal meth, methamphetamines, cocaine) within 60 days prior to randomization.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-07-12 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness. | 24 and 48 weeks.
  Effectiveness: Individuals with >50 copies/ml.
Safety of switching ART regimen with an INSTI to DTG/3TC. | 24 and 48 weeks.
  Number of participants with treatment-related adverse events as assessed of serious adverse events (WHO grade 3 or 4) for PWH treated with DTG/3TC at 24 and 48 weeks, expressed in proportions of new cases.
Tolerability of switching ART regimen with an INSTI to DTG/3TC. | 24 and 48 weeks.
  Maintaining ART with DTG/3TC without changes, interruptions, or substitutions due to adverse effects or perceived discomfort.

SECONDARY OUTCOMES:
Changes in lipid profile. | 24 and 48 weeks
  Changes in total cholesterol, HDL cholesterol, and triglycerides, measured in mg/dL.
Changes in body mass index | 24 and 48 weeks.
  To evaluate changes in body mass index (BMI, kg/m²) at weeks 24 and 48.
Changes in waist circumference. | 24 and 48 weeks.
  To evaluate changes greater than 90 cm in waist circumference at weeks 24 and 48.
Glucose metabolism disorders. | 24 and 48 weeks.
  To determine changes at weeks 24 and 48, including the development of prediabetes or diabetes.
Assess changes in blood pressure and cardiovascular risk | 24 and 48 weeks
  Framingham and AHA/ACC scales
Measure body composition | 24 and 48 weeks
  fat, water, muscle

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Infectología, Centro Médico Nacional La Raza, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
The data cannot be shared openly because it contains personal information about the participants; if required, it can be requested from the corresponding author.

REFERENCES:
- [Background] MacPherson DW, Gushulak BD. Human mobility and population health. New approaches in a globalizing world. Perspect Biol Med. 2001 Summer;44(3):390-401. doi: 10.1353/pbm.2001.0053. PMID 11482008
- [Background] Mann RB, Solodukhin SN. Conical geometry and quantum entropy of a charged Kerr black hole. Phys Rev D Part Fields. 1996 Sep 15;54(6):3932-3940. doi: 10.1103/physrevd.54.3932. No abstract available. PMID 10021070
- [Background] Venkiteswaran K, Sgoutas DS, Santanam N, Neylan JF. Tacrolimus, cyclosporine and plasma lipoproteins in renal transplant recipients. Transpl Int. 2001 Dec;14(6):405-10. doi: 10.1007/s001470100006. PMID 11793038
- [Background] van Wyk J, Ajana F, Bisshop F, De Wit S, Osiyemi O, Portilla Sogorb J, Routy JP, Wyen C, Ait-Khaled M, Nascimento MC, Pappa KA, Wang R, Wright J, Tenorio AR, Wynne B, Aboud M, Gartland MJ, Smith KY. Efficacy and Safety of Switching to Dolutegravir/Lamivudine Fixed-Dose 2-Drug Regimen vs Continuing a Tenofovir Alafenamide-Based 3- or 4-Drug Regimen for Maintenance of Virologic Suppression in Adults Living With Human Immunodeficiency Virus Type 1: Phase 3, Randomized, Noninferiority TANGO Study. Clin Infect Dis. 2020 Nov 5;71(8):1920-1929. doi: 10.1093/cid/ciz1243. PMID 31905383